CLINICAL TRIAL: NCT06726109
Title: a FOCUSed Prospective Registry on Acute Decompensation of Heart Failure With Reduced Ejection Fraction- The FOCUS-ADHF Registry
Brief Title: The FOCUS-ADHF Registry
Acronym: FOCUS-ADHF
Status: Recruiting | Type: Observational
Sponsor: ASL Città di Torino (Other)
Collaborators: Hospital of Rivoli (Unknown); Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Maurizio Bertaina, Medical Doctor, Principal Investigator, Ospedale S. Giovanni Bosco
Other Study IDs: 01
Record Dates: First submitted 2024-11-20; First posted 2024-12-10 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Acute Heart Failure With Reduced Ejection Fraction; Decompensation; Heart, Congestive; Regurgitation, Mitral
Keywords: Acute Heart Failure (AHF); Acute Decompensated Heart Failure (ADHF); Vasodilators; Dilated left ventricle; reduced ejection fraction (rEF); functional mitral regurgitation (FMR); increased filling pressure; increased pulmonary artery pressure; nitroprusside; sodium nitroprusside; Isosorbide Dinitrate; nitroglycerine
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- vasodilator treated: patients treated with vasodilator therapy after admission for an ADHF episode
- Not vasodilator treated: Patients not treated with vasodilator therapy after admission for an ADHF episode

SUMMARY:
Acute heart failure (AHF) represents a significant clinical and economic burden due to its impact on patients' quality of life, poor prognosis, and high healthcare costs. Despite advancements in treatment, the optimal therapeutic management of these patients, particularly those with severely reduced ejection fraction and dilated left ventricles, remains uncertain. The last European Society of Cardiology (ESC) guidelines gave a weak recommendation for using intravenous (IV) vasodilators in patients with adequate systolic blood pressure. This is derived from heterogeneous randomized controlled trials (RCTs) enrolling all-comers heart failure patients. Those studies did not specifically target conditions that from a pathophysiological perspective might derive potential positive response from vasodilators like left ventricle dilatation, significant mitral regurgitation and/or increased filling pressure. Patients with such characteristics show higher myocardial wall tension and are particularly vulnerable to afterload increases, positioning them as optimal candidates for vasodilator therapy during acute decompensation. Little evidence is available from real world cohort study on the benefit of vasodilators in this group of patients. Many of these studies used pre-defined protocol and invasive hemodynamic monitoring. On the contrary the use of echocardiographic evaluation to phenotype, infer hemodynamic parameters and assess treatment effect has become the most common adopted technique in real life.

The present prospective registry aims to investigate acute treatment management and outcomes in a focused population of patients admitted for an acute decompensation of heart failure (ADHF) with severely reduced ejection fraction and dilated left ventricle or significant functional mitral regurgitation.

Inclusion Criteria:

* Patients within 24h since admission for an ADHF defined as

  1. signs and symptoms of volume overload with necessity of iv diuretic treatment.
  2. and NT-proBNP (N-terminal pro-B-type natriuretic peptide) >1500 pg/mL or a B-type natriuretic peptide level of >500 ng/mL.

     • Admission echocardiography with evidence of a dilated left ventricle and/or at least moderate functional mitral regurgitation (FMR), reduced ejection fraction (<40%), increased LV (II/III degree diastolic dysfunction) and pulmonary pressure (sPAP ≥ 40 mmHg or MPAP ≥ 20 mmHg).

     Exclusion Criteria:

     - Cardiogenic shock at admission warranting immediate MCS / inotropic support, severe renal or hepatic impairment, recent myocardial infarction, and other terminal illnesses.
     * Use of vasopressors/inotropes or mechanical support at admission. Methods Patients will receive treatments according to their physician's discretion based on ESC guidelines. Serial evaluations of heart function will be conducted using echocardiography and lung ultrasound (LUS) at multiple time points as well as hemodynamic data, laboratory and HF medications' prescription and dosages Primary endpoint

       * 3 months incidence of need of Heart Replacement Therapies (LVAD or heart transplantation) and/or heart failure re-hospitalization and/or all-cause death.

     Secondary endpoints • In hospital and 3 months All-cause death

     • All cause and HF related hospitalizations within 3 months

     • Heart replacement therapies (LVAD or heart transplantation) within 3 months.

     • In hospital Worsening Heart Failure (WHF)

     • Need of renal replacement therapy (RRT) within 3 months

     • In-hospital length of stay (days), NT-proBNP variations, GDMT and diuretics prescription and dosages up to three months;

     Objectives:

  <!-- -->

  1. To describe the acute therapeutic management and discharge prescriptions for heart failure medications, including doses, in a selected population with ADHF.
  2. To evaluate clinical outcomes and NT-proBNP variation in relation to initial intravenous medications, particularly comparing the use versus non-use of vasodilators.
  3. To identify the incidence and timing of a significant therapeutic response through serial evaluations of LUS and echo-derived parameters, and to examine their association with the initial intravenous medications prescribed.
  4. To investigate the association between the criteria for therapeutic response and clinical outcomes in both short- and medium-term follow-up, with a focus on the relationship to the initially administered therapy.

DETAILED DESCRIPTION:
This is a real-life, observational, prospective multicenter registry. Patients fulfilling inclusion and exclusion criteria will be consecutively enrolled in enrolling center.

Enrolled patients will be treated at each treating physician's discretion referring to the general recommendation of the last ESC guidelines on management of acute heart failure as well as local practice. General guidelines for vasodilators use will be shared among enrolling centers to increase uniformity of treatment in case of prescription of this strategy.

-After achievement of adequate decongestion, iv vasodilators infusion (if used) will be weaned and HF medications introduction/titration up to guidelines recommended doses.

Other therapeutic interventions: will be left to treating physician discretion aiming to decongest the patient.

Starting inotropes, vasopressors, mechanical cardiac support device (MCS) and use of non-invasive and/or invasive ventilation as well as continuous renal replacement therapies (CRRT) will be left to the treating physicians' discretion according to clinical course.

ELIGIBILITY:
Inclusion Criteria:

* Patients within 24h since admission for an acute decompensation of heart failure (ADHF)* (both acute on chronic and de novo) defined as

  1. signs and symptoms of volume overload with necessity of iv diuretic treatment.
  2. and NT-proBNP (N-terminal pro-B-type natriuretic peptide) >1500 pg/mL or a B-type natriuretic peptide level of >500 ng/mL.

AND ALL THE FOLLOWING echo entry criteria at admission:

1. A dilated left ventricle (defined as a indexed LVEDD ≥ 31 mm/sm and ≥ 32 mm/sm or a indexed LVEDVol ≥ 75 ml/sm and ≥ 62 ml/sm in men and women respectively) AND/OR at least moderate functional mitral regurgitation (FMR).
2. Reduced ejection fraction (<40%)
3. Increased LV filling pressure (defined as II°-III° Diastolic dysfunction) AND increased pulmonary artery pressure (i.e. echo estimated systolic pulmonary artery pressure [sPAP] ≥ 40 mmhg and/or echo estimated mean pulmonary artery pressure [mPAP] ≥ 20 mmHg).

Exclusion Criteria:

* Patients presenting in Cardiogenic shock defined as hypotension (SBP < 90mmHg or MAP ≤ 55) AND hypoperfusion (defined as arterial lactates > 4 mmol/L)
* Estimated GFR <=20 ml/min/1.73 m2 or in chronic renal replacement therapies.
* End-stage hepatic impairment
* Use of temporary mechanical support at the moment of study inclusion or planned to use it within hours (IABP; Impella, VA ECMO)
* Ongoing treatment with vasopressors/inotropes at the moment of randomization or administration of Levosimendan within 30 days before randomization. Patients admitted for a planned cycle of Levosimendan infusion will be excluded by the present study as well.
* AHF secondary to recent onset tachy-arrhythmias
* ST tract elevated myocardial infarction (STEMI) < 30 days, myocarditis <30 days, AHF due to severe primary valve disease or clinical suspicion of an acute mechanical cause of AHF
* restrictive cardiomyopathy, constrictive pericarditis, hypertrophic obstructive cardiomyopathy, tako-tsubo syndrome
* Infective endocarditis, concomitant active septic disease as predominant cause of decompensation or admission TC>38°c.
* LVAD carriers or Heart transplant recipients
* Terminal illness other than heart failure with an expected survival <180 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All-comers patients admitted for an ADHF with a severely reduced ejection fraction, a dilated left ventricle or significant functional mitral regurgitation (FMR) and increased left ventricle filling and pulmonary pressures as estimated by echocardiographic evaluation at admission.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-04-27 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
incidence of need of Heart Replacement Therapies (LVAD or heart transplantation) and/or heart failure re-hospitalization and/or all-cause death. | from enrollment up to 3 months

SECONDARY OUTCOMES:
incidence of all-cause mortality | from enrollment up to 3 months
incidence of HF related hospitalizations | from enrollment up to 3 months
incidence of all-cause hospitalization | from enrollment up to 3 months
incidence of patients needing heart replacement therapies (LVAD or heart transplantation) | from enrollment up to 3 months
  Heart transplantation or LVAD implantation
incidence of In hospital Worsening Heart Failure (WHF) | from date of enrollment until the date of first worsening heart failure event or the date of death from any cause or the date of hospital discharge, whichever came first, assessed up to 3 months
  need for therapeutic intensification for inadequate clinical response
incidence of patients needing renal replacement therapy (RRT) | from enrollment up to 3 months
  need for use of renal replacement therapy
rate of GDMT and diuretics prescription and dosages | from admission up to 3 months follow-up
  prescription of 4 hf pillars, Vericiguat, diuretics and doses

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Bertaina, MD, Principal Investigator — Division of Cardiology, San Giovanni Bosco,ASL Città di Torino, Turin, Italy; Wilfred Mullens, MD,Prof., Principal Investigator — Division of Cardiology,Ziekenhuis Oost-Limburg, Genk, Belgium. Hasselt University, Belgium.; Alessandro Galluzzo, MD, Principal Investigator — Division of cardiology, Rivoli Hospital, Rivoli, Italy
Locations (4):
- division of Cardiology, Ziekenhuis Oost-Limburg, Genk, Belgium. Hasselt University, Belgium., Genk, Belgium, Belgium
- Italy (3):
  - Rivoli Hospital, Rivoli, Italy
  - San Giovanni Bosco Hospital, Turin, Italy
  - Santa Maria della Misericordia, Azienda sanitaria universitaria Friuli Centrale,, Udine, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Platz E, Jhund PS, Girerd N, Pivetta E, McMurray JJV, Peacock WF, Masip J, Martin-Sanchez FJ, Miro O, Price S, Cullen L, Maisel AS, Vrints C, Cowie MR, DiSomma S, Bueno H, Mebazaa A, Gualandro DM, Tavares M, Metra M, Coats AJS, Ruschitzka F, Seferovic PM, Mueller C; Study Group on Acute Heart Failure of the Acute Cardiovascular Care Association and the Heart Failure Association of the European Society of Cardiology. Expert consensus document: Reporting checklist for quantification of pulmonary congestion by lung ultrasound in heart failure. Eur J Heart Fail. 2019 Jul;21(7):844-851. doi: 10.1002/ejhf.1499. Epub 2019 Jun 19. PMID 31218825
- [Background] Metra M, Adamo M, Tomasoni D, Mebazaa A, Bayes-Genis A, Abdelhamid M, Adamopoulos S, Anker SD, Bauersachs J, Belenkov Y, Bohm M, Gal TB, Butler J, Cohen-Solal A, Filippatos G, Gustafsson F, Hill L, Jaarsma T, Jankowska EA, Lainscak M, Lopatin Y, Lund LH, McDonagh T, Milicic D, Moura B, Mullens W, Piepoli M, Polovina M, Ponikowski P, Rakisheva A, Ristic A, Savarese G, Seferovic P, Sharma R, Thum T, Tocchetti CG, Van Linthout S, Vitale C, Von Haehling S, Volterrani M, Coats AJS, Chioncel O, Rosano G. Pre-discharge and early post-discharge management of patients hospitalized for acute heart failure: A scientific statement by the Heart Failure Association of the ESC. Eur J Heart Fail. 2023 Jul;25(7):1115-1131. doi: 10.1002/ejhf.2888. Epub 2023 Jul 13. PMID 37448210
- [Background] Gentile F, Buoncristiani F, Sciarrone P, Bazan L, Panichella G, Gasparini S, Chubuchny V, Taddei C, Poggianti E, Fabiani I, Petersen C, Lancellotti P, Passino C, Emdin M, Giannoni A. Left ventricular outflow tract velocity-time integral improves outcome prediction in patients with secondary mitral regurgitation. Int J Cardiol. 2023 Dec 1;392:131272. doi: 10.1016/j.ijcard.2023.131272. Epub 2023 Aug 19. PMID 37604287
- [Background] Frea S, Gravinese C, Boretto P, De Lio G, Bocchino PP, Angelini F, Cingolani M, Gallone G, Montefusco A, Valente E, Pidello S, Raineri C, De Ferrari GM. Comprehensive non-invasive haemodynamic assessment in acute decompensated heart failure-related cardiogenic shock: a step towards echodynamics. Eur Heart J Acute Cardiovasc Care. 2024 Sep 25;13(9):646-655. doi: 10.1093/ehjacc/zuae087. PMID 39012797
- [Background] Bertaina M, Galluzzo A, Rossello X, Sbarra P, Petitti E, Prever SB, Boccuzzi G, D'Ascenzo F, Frea S, Pidello S, Morici N, Sacco A, Oliva F, Valente S, De Ferrari GM, Ugo F, Rametta F, Attisani M, Zanini P, Noussan P, Iannaccone M. Prognostic implications of pulmonary artery catheter monitoring in patients with cardiogenic shock: A systematic review and meta-analysis of observational studies. J Crit Care. 2022 Jun;69:154024. doi: 10.1016/j.jcrc.2022.154024. Epub 2022 Mar 25. PMID 35344825
- [Background] Hill JA, Pauly DF, Olitsky DR, Russell S, O'Connor CM, Patterson B, Elkayam U, Khan S, Stevenson LW, Brooks K, Wagoner L, Conway G, Koelling T, Huysen C Van, Hare J, Breton E, Adams KF, Glotzer J, Fonarow G, Hamilton M, Sorg J, Drazner M, Hoffman S, Miller LW, Graziano JA, Berman ME, Frantz R, Hartman K, Leier C V., Abraham WT, et al. Evaluation study of congestive heart failure and pulmonary artery catheterization effectiveness. J Am Med Assoc 2005;294:1625-1633.
- [Background] Verbrugge FH, Dupont M, Finucan M, Gabi A, Hawwa N, Mullens W, Taylor DO, Young JB, Starling RC, Tang WH. Response and tolerance to oral vasodilator up-titration after intravenous vasodilator therapy in advanced decompensated heart failure. Eur J Heart Fail. 2015 Sep;17(9):956-63. doi: 10.1002/ejhf.324. Epub 2015 Jul 24. PMID 26213182
- [Background] Mullens W, Abrahams Z, Francis GS, Skouri HN, Starling RC, Young JB, Taylor DO, Tang WH. Sodium nitroprusside for advanced low-output heart failure. J Am Coll Cardiol. 2008 Jul 15;52(3):200-7. doi: 10.1016/j.jacc.2008.02.083. PMID 18617068
- [Background] Garatti L, Frea S, Bocchino PP, Angelini F, Cingolani M, Sacco A, Rondinara GM, Bagnardi V, Sala IM, Kapur NK, Colombo PC, De Ferrari GM, Morici N. Sodium nitroprusside in acute heart failure: A multicenter historic cohort study. Int J Cardiol. 2022 Dec 15;369:37-44. doi: 10.1016/j.ijcard.2022.08.009. Epub 2022 Aug 6. PMID 35944767
- [Background] Freund Y, Cachanado M, Delannoy Q, Laribi S, Yordanov Y, Gorlicki J, Chouihed T, Feral-Pierssens AL, Truchot J, Desmettre T, Occelli C, Bobbia X, Khellaf M, Ganansia O, Bokobza J, Balen F, Beaune S, Bloom B, Simon T, Mebazaa A. Effect of an Emergency Department Care Bundle on 30-Day Hospital Discharge and Survival Among Elderly Patients With Acute Heart Failure: The ELISABETH Randomized Clinical Trial. JAMA. 2020 Nov 17;324(19):1948-1956. doi: 10.1001/jama.2020.19378. PMID 33201202
- [Background] Kozhuharov N, Goudev A, Flores D, Maeder MT, Walter J, Shrestha S, Gualandro DM, de Oliveira Junior MT, Sabti Z, Muller B, Noveanu M, Socrates T, Ziller R, Bayes-Genis A, Sionis A, Simon P, Michou E, Gujer S, Gori T, Wenzel P, Pfister O, Conen D, Kapos I, Kobza R, Rickli H, Breidthardt T, Munzel T, Erne P, Mueller C; GALACTIC Investigators; Mueller C, Erne P, Muller B, Rickli H, Maeder M, Tavares de Oliveira M Jr, Munzel T, Bayes-Genis A, Sionis A, Goudev A, Dimov B, Hartwiger S, Arenja N, Glatz B, Herr N, Isenrich R, Mosimann T, Twerenbold R, Boeddinghaus J, Nestelberger T, Puelacher C, Freese M, Vogele J, Meissner K, Martin J, Strebel I, Wussler D, Schumacher C, Osswald S, Vogt F, Hilti J, Barata S, Schneider D, Schwarz J, Fitze B, Hartwiger S, Arenja N, Glatz B, Herr N, Isenrich R, Mosimann T, Twerenbold R, Boeddinghaus J, Nestelberger T, Puelacher C, Freese M, Vogele J, Meissner K, Martin J, Strebel I, Wussler D, Schumacher C, Osswald S, Vogt F, Hilti J, Barata S, Schneider D, Schwarz J, Fitze B, Arenja N, Rentsch K, Bossa A, Jallad S, Soeiro A, Georgiev D, Jansen T, Gebel G, Bossard M, Christ M. Effect of a Strategy of Comprehensive Vasodilation vs Usual Care on Mortality and Heart Failure Rehospitalization Among Patients With Acute Heart Failure: The GALACTIC Randomized Clinical Trial. JAMA. 2019 Dec 17;322(23):2292-2302. doi: 10.1001/jama.2019.18598. PMID 31846016
- [Background] Metra M, Teerlink JR, Cotter G, Davison BA, Felker GM, Filippatos G, Greenberg BH, Pang PS, Ponikowski P, Voors AA, Adams KF, Anker SD, Arias-Mendoza A, Avendaño P, Bacal F, Böhm M, Bortman G, Cleland JGF, Cohen-Solal A, Crespo-Leiro MG, Dorobantu M, Echeverría LE, Ferrari R, Goland S, Goncalvesová E, Goudev A, Køber L, Lema-Osores J, Levy PD, McDonald K, et al. Effects of Serelaxin in Patients with Acute Heart Failure. N Engl J Med N Engl J Med; 2019;381:716-726.
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, González-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, Meer P Van Der, Sisakian HS, Isayev E, Kurlianskaya A, Mullens W, Tokmakova M, Agathangelou P, Melenovsky V, Wiggers H, Hassanein M, et al. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J 2016;37:2129-2200m.
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Böhm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J Oxford Academic; 2021;42:3599-3726.